CLINICAL TRIAL: NCT03246152
Title: Evaluation of the Effect of Repeated Intravitreal Injections of Anti-VEGF on Macular Perfusion in Diabetic Patients Using Optical Coherence Tomography Angiography
Brief Title: Evaluation of the Effect of Intravitreal Injections of Anti-VEGF on Macular Perfusion in Diabetic Patients Using OCTA
Acronym: IMPACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Gehad Elnahry, Clinical Demonstrator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-79-2017
Record Dates: First submitted 2017-08-06; First posted 2017-08-11 (Actual); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Macular Edema; Ischemic Maculopathy
Keywords: Anti-VEGF safety; Ischemic Maculopathy; Diabetic Macular Edema; OCTA
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bevacizumab group (Experimental): Monthly intravitreal injection of 2.5 mg of Bevacizumab for at least 3 consecutive months. This is followed by treat and extend regimen after resolution of macular edema.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Repeated intravitreal injections of Bevacizumab monthly
  Other Names: Avastin

SUMMARY:
Anti-vascular endothelial growth factor (VEGF) drugs are the mainstay of therapy for diabetic macular edema (DME), substantially improving visual acuity for many diabetics worldwide, and proving effective for treatment of both non-proliferative and proliferative diabetic retinopathy.

Many studies such as Diabetic Retinopathy Clinical Research Network studies, RESTORE Study, and The BOLT Study have supported the use of different anti-VEGF agents in the treatment of DME with better visual outcomes using anti-VEGF injections alone or in combination with other treatments.

Several ocular complications of intravitreal anti-VEGF injections have been reported including endophthalmitis, cataract and retinal detachment. The effect of anti-VEGF drugs on macular perfusion has been inconclusive, with mixed reports of increase, decrease or no effect on perfusion in response to anti-VEGF treatment. In many of these studies, however, patients with more ischaemic retinas were not included. Retinal ischemia is an important factor in the progression and prognosis of diabetic retinopathy.

Fluorescein angiography (FA) was the method used to assess changes in macular perfusion after anti-VEGF injections in most of the studies. Despite its clinical usefulness, however, FA is known to have documented risks. Optical coherence tomography angiography (OCTA) is a new noninvasive method of acquiring high-resolution images of the retinal vasculature that can be utilized in the treatment of retinal disease without the need for dye injection. It allows the visualization of the superficial and deep retinal capillary layers separately and the construction of microvascular flow maps.

Several studies have proved the reliability of OCTA in detecting and quantifying macular ischemia in diabetics.

In this study, investigators aim to evaluate the effect of repeated intravitreal injections of different Anti-VEGF agents on the perfusion of different capillary layers in the macula of diabetic patients using OCTA.

DETAILED DESCRIPTION:
This is a prospective interventional study to evaluate the effect of repeated intravitreal injections of Anti-VEGF on macular perfusion in diabetic patients using optical coherence tomography angiography (OCTA).

Each patient will receive a detailed ophthalmologic examination including measurement of BCVA as well as applanation tonometry, undilated and dilated slit-lamp biomicroscopic examination and indirect fundus examination.

Duration of diabetes and its control through HbA1C measurement will be recorded for each patient.

Type 1 and 2 diabetic patients found to have BCVA worse than 6/6 and clinical evidence of macular edema will undergo SD OCT and FA.

Patients with center involved macula edema detected by SD OCT will be included in the study and will undergo baseline macular OCTA.

These patients will then undergo intravitreal injections of Anti-VEGF monthly for 3 months then OCTA will be repeated to evaluate changes in macular perfusion and SD OCT will be repeated to assess retinal thickness. Patients with center involving macular edema on SD-OCT after the first 3 injections will continue to receive intravitreal Anti-VEGF injections monthly until the edema subsides or the study duration ends. These patients then undergo a final macular OCTA for perfusion evaluation and SD OCT for thickness assessment.

OCTA will be performed with an Avanti RTVue XR system (Optovue, Inc., Fremont, CA, USA). Area of FAZ and capillary density at each capillary layer will be calculated before and after interventions using the OCTA machine software and ImageJ software.

All statistical analyses will be done using IBM SPSS v20.0 statistical software (IBM Corporation, NY, USA). Descriptive statistics will be calculated, and the data will be summarized as mean ± SD for numerical data, and as frequencies and percentages for categorical data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Type 1 or 2 diabetes mellitus
3. Decreased BCVA due to diabetic macular edema
4. Center involvement by the edema on spectral domain optical coherence tomography (SD OCT)
5. Any stage of diabetic retinopathy

Exclusion Criteria:

1. Ocular conditions that may affect macular perfusion (e.g. retinal vascular diseases, uveitis, vasculitis etc.)
2. History of vitreoretinal surgeries (excluding intravitreal injections)
3. Any previous treatment for diabetic macular edema
4. Presence of epiretinal membrane involving the macula or vitreomacular traction
5. Media opacity preventing good image quality
6. Uncontrolled glaucoma
7. Thromboembolic events within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled E El Rakhawy, PhD, Study Director — Cairo University; Karim A Raafat, PhD, Study Director — Cairo University; Ahmed AA Abdel Kader, PhD, Study Chair — Cairo University; Ayman GA Elnahry, MSc, Principal Investigator — Cairo University
Locations (1):
- Cairo University Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajlan RS, Silva PS, Sun JK. Vascular Endothelial Growth Factor and Diabetic Retinal Disease. Semin Ophthalmol. 2016;31(1-2):40-8. doi: 10.3109/08820538.2015.1114833. PMID 26959128
- [Background] Michaelides M, Kaines A, Hamilton RD, Fraser-Bell S, Rajendram R, Quhill F, Boos CJ, Xing W, Egan C, Peto T, Bunce C, Leslie RD, Hykin PG. A prospective randomized trial of intravitreal bevacizumab or laser therapy in the management of diabetic macular edema (BOLT study) 12-month data: report 2. Ophthalmology. 2010 Jun;117(6):1078-1086.e2. doi: 10.1016/j.ophtha.2010.03.045. Epub 2010 Apr 22. PMID 20416952
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Avery RL. Regression of retinal and iris neovascularization after intravitreal bevacizumab (Avastin) treatment. Retina. 2006 Mar;26(3):352-4. doi: 10.1097/00006982-200603000-00016. No abstract available. PMID 16508438
- [Background] Chapman JA, Beckey C. Pegaptanib: a novel approach to ocular neovascularization. Ann Pharmacother. 2006 Jul-Aug;40(7-8):1322-6. doi: 10.1345/aph.1G604. Epub 2006 Jul 18. PMID 16849623
- [Background] Zhang X, Bao S, Hambly BD, Gillies MC. Vascular endothelial growth factor-A: a multifunctional molecular player in diabetic retinopathy. Int J Biochem Cell Biol. 2009 Dec;41(12):2368-71. doi: 10.1016/j.biocel.2009.07.011. Epub 2009 Jul 29. PMID 19646547
- [Background] Hwang TS, Gao SS, Liu L, Lauer AK, Bailey ST, Flaxel CJ, Wilson DJ, Huang D, Jia Y. Automated Quantification of Capillary Nonperfusion Using Optical Coherence Tomography Angiography in Diabetic Retinopathy. JAMA Ophthalmol. 2016 Apr;134(4):367-73. doi: 10.1001/jamaophthalmol.2015.5658. PMID 26795548
- [Background] Bradley PD, Sim DA, Keane PA, Cardoso J, Agrawal R, Tufail A, Egan CA. The Evaluation of Diabetic Macular Ischemia Using Optical Coherence Tomography Angiography. Invest Ophthalmol Vis Sci. 2016 Feb;57(2):626-31. doi: 10.1167/iovs.15-18034. PMID 26903223
- [Background] Freiberg FJ, Pfau M, Wons J, Wirth MA, Becker MD, Michels S. Optical coherence tomography angiography of the foveal avascular zone in diabetic retinopathy. Graefes Arch Clin Exp Ophthalmol. 2016 Jun;254(6):1051-8. doi: 10.1007/s00417-015-3148-2. Epub 2015 Sep 4. PMID 26338819
- [Background] Spaide RF, Klancnik JM Jr, Cooney MJ. Retinal vascular layers imaged by fluorescein angiography and optical coherence tomography angiography. JAMA Ophthalmol. 2015 Jan;133(1):45-50. doi: 10.1001/jamaophthalmol.2014.3616. PMID 25317632
- [Background] Yannuzzi LA, Rohrer KT, Tindel LJ, Sobel RS, Costanza MA, Shields W, Zang E. Fluorescein angiography complication survey. Ophthalmology. 1986 May;93(5):611-7. doi: 10.1016/s0161-6420(86)33697-2. PMID 3523356
- [Background] Bonnin P, Pournaras JA, Lazrak Z, Cohen SY, Legargasson JF, Gaudric A, Levy BI, Massin P. Ultrasound assessment of short-term ocular vascular effects of intravitreal injection of bevacizumab (Avastin((R)) ) in neovascular age-related macular degeneration. Acta Ophthalmol. 2010 Sep;88(6):641-5. doi: 10.1111/j.1755-3768.2009.01526.x. PMID 19563370
- [Background] Papadopoulou DN, Mendrinos E, Mangioris G, Donati G, Pournaras CJ. Intravitreal ranibizumab may induce retinal arteriolar vasoconstriction in patients with neovascular age-related macular degeneration. Ophthalmology. 2009 Sep;116(9):1755-61. doi: 10.1016/j.ophtha.2009.03.017. Epub 2009 Jun 27. PMID 19560206
- [Background] Manousaridis K, Talks J. Macular ischaemia: a contraindication for anti-VEGF treatment in retinal vascular disease? Br J Ophthalmol. 2012 Feb;96(2):179-84. doi: 10.1136/bjophthalmol-2011-301087. PMID 22250209
- [Background] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Background] Mitchell P, Bandello F, Schmidt-Erfurth U, Lang GE, Massin P, Schlingemann RO, Sutter F, Simader C, Burian G, Gerstner O, Weichselberger A; RESTORE study group. The RESTORE study: ranibizumab monotherapy or combined with laser versus laser monotherapy for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):615-25. doi: 10.1016/j.ophtha.2011.01.031. PMID 21459215
- [Derived] Elnahry AG, Abdel-Kader AA, Raafat KA, Elrakhawy K. Evaluation of Changes in Macular Perfusion Detected by Optical Coherence Tomography Angiography following 3 Intravitreal Monthly Bevacizumab Injections for Diabetic Macular Edema in the IMPACT Study. J Ophthalmol. 2020 Apr 27;2020:5814165. doi: 10.1155/2020/5814165. eCollection 2020. PMID 32411431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is the number of enrolled patients that completed the study.
Groups:
- Bevacizumab Group: Monthly intravitreal injection of Bevacizumab for at least 3 consecutive months. This is followed by treat and extend regimen after resolution of macular edema.
  Bevacizumab: Repeated intravitreal injections of Bevacizumab monthly
Period: Overall Study
Arm/Group | Bevacizumab Group
Started | 31
Completed | 28
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab Group
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 31
Region of Enrollment [Number; unit: participants]
  Egypt | 31

OUTCOME MEASURES:

1. Primary Outcome: FAZ Area Change
Description: Effect of repeated intravitreal Anti-VEGF injections on Foveal Avascular Zone (FAZ) area measured using the freehand tool of ImageJ
Time Frame: At baseline and after 3-6 consecutive monthly injections.
Population: Patients with adequate image quality
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Bevacizumab Group
Number analyzed (Participants) | 26
mm^2 | 0.03 (0.1)

2. Primary Outcome: Macular Capillary Density Change at Full Retinal Thickness
Description: Effect of repeated intravitreal Anti-VEGF injections on macular capillary density using the change in the skeletonized vascular density and fractal dimension measured by ImageJ
Time Frame: At baseline and after 3-6 consecutive monthly injections.
Population: Patients with adequate image quality
Measure: Mean (Standard Deviation); unit: percentage of vascularity
Arm/Group | Bevacizumab Group
Number analyzed (Participants) | 26
percentage of vascularity | -2.5 (5.72)

3. Secondary Outcome: BCVA Change
Description: Correlation of BCVA change with degree of capillary non-perfusion before and after injections
Time Frame: At baseline and after 3-6 consecutive monthly injections.
Population: Patients with good image quality
Measure: Mean (Standard Deviation); unit: Logmar
Arm/Group | Bevacizumab Group
Number analyzed (Participants) | 26
Logmar | -0.21 (0.27)
Statistical Analysis 1: Comparison: Bevacizumab Group; Correlation between change in BCVA and the pre treatment, post treatment, and change in vascular density following 3-6 injections was performed; Test type: Other; p > 0.05, Pearson's correlation coefficient

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Bevacizumab Group
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 18/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Group (N=31)
Subconjunctival hemorrhage (Eye disorders) | 13
Ocular irritation (Eye disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03246152/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT03246152/SAP_001.pdf